CLINICAL TRIAL: NCT06634004
Title: Personalized Hemodynamic and Metabolic Signatures of Revascularization Response in Moyamoya Disease
Brief Title: Biomarker-Led Optimization of Successful Surgical Outcomes in Moyamoya
Acronym: BLOSSOM
Status: Enrolling by invitation | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Manus Donahue, Professor of Neurology, Vanderbilt University Medical Center
Other Study IDs: 231114; 1R01NS133101 (NIH)
Record Dates: First submitted 2024-09-30; First posted 2024-10-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Moyamoya Disease
Keywords: moyamoya; stroke
MeSH Terms: conditions — Moyamoya Disease; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (10 mL) and Urine (10 mL) samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Moyamoya: Adults diagnosed with Moyamoya who are being considered for revascularization surgery.
  Interventions: Other: BOLD MRI
- Control: Healthy adults who will under go a BOLD MRI for research purposes.
  Interventions: Other: BOLD MRI

INTERVENTIONS:
Other: BOLD MRI — The study will utilize the MRI diagnostic reactivity test to evaluate cerebrovascular reactivity in patients with moyamoya and healthy controls. All participants (patients and controls) receive the same diagnostic scan, and there is no cross-over, factorial, or sequential nature to the study.

SUMMARY:
The goal of this work is to use advanced magnetic resonance imaging (MRI) methods to assess brain blood flow and vascular function in adults with moyamoya disease (MMD). MMD is a condition characterized by narrowing or obstruction of major arteries in the brain and people with MMD have a high risk of stroke. Study participants will be enrolled from Vanderbilt University Medical Center and Johns Hopkins Hospital and will undergo up to two MRI scans where measurements of cerebrovascular reserve are performed using inhaled room air mixed with 5% carbon dioxide. Scans will be performed before and after surgeries to treat MMD, all surgeries are clinically indicated and are not research procedures. To further understand how surgeries impact brain health, we will also perform neurological exams and cognitive testing at approximately the same time as the imaging scans. The overall goal is to incorporate advanced imaging and cognitive assessments to understand how surgeries improve brain health in these patients, and furthermore, to use this information to develop improved screening tools for stroke risk and decisions about surgery.

DETAILED DESCRIPTION:
MMD is a condition with narrowing and blockage of major arteries in the brain and people with MMD have a high risk of stroke. Neurosurgical revascularization surgery is usually recommended to provide more blood flow to the brain and hopefully prevent further strokes. The primary goal of this study to improve the understanding of response to neurosurgical treatment and disease improvement or progression by using innovative magnetic resonance imaging (MRI) methods to assess brain blood flow and oxygen use in adults with idiopathic MMD before and after they have surgery.

The study will recruit 100 adults with idiopathic MMD, aged 18-60 years, from neurosurgery clinics at Vanderbilt University Medical Center and Johns Hopkins Hospital, as well as 20 healthy controls. Participants will undergo comprehensive evaluations including MRI, cognitive exams, and optional blood and urine collection.

More specifically, the proposal involves the development and application of MRI methods for visualizing hemodynamic and metabolic relationships in adults suffering from idiopathic moyamoya disease. As part of the research study, participants will undergo 1-2 MRI scans at a field strength of 3 Tesla. Each scan session will last approximately one hour, which will include the time when the volunteers rehearse the experiment outside of the scanner, time for the volunteers to be comfortably placed in the scanner, scanning (including one scan where blood flow and oxygenation will be measured before and during a mild hypercapnic stimulus), and finally time for the participants to slowly exit the scan room. Moyamoya participants may also undergo surgical revascularization and catheter angiography using digital subtraction angiography (DSA). These procedures are clinically indicated and will be performed as part of clinical care, and therefore are not research procedures. Therefore, the risks relevant to this study pertain to the research procedures only, which are comprised of non-invasive MRI scans, neurological exams, as well as cognitive testing. Neurological assessments will utilize the NIH Stroke Scale (NIHSS) and the modified Rankin Score (mRS) to evaluate disability. Neurocognitive testing will be completed to assess multiple cognitive domains.

Participants are not randomized to an intervention or study group but studying cerebral blood flow changes is considered a basic experimental study involving humans (BESH) clinical trial by the National Institutes of Health that funds this study. The study uses commercial MRI approaches and data-driven software approaches to ensure the tools are generalizable across medical centers. This comprehensive approach aims to identify which patients require specific treatments and understand what contributes to positive responses. Planned surgery for MMD is an inclusion criteria for this study for MMD participants. Again, surgery will be performed as a part of clinical care and is not a research procedure. Therefore, the risks relevant to this study pertain to the research procedures only, which are comprised of non-invasive MRI scans, neurological exams, as well as cognitive testing, blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

Moyamoya

1. Clinical diagnosis of moyamoya disease as defined by gold-standard catheter angiography and consensus adjudication of imaging and neurological findings
2. Age = 18-60 years
3. Participants for the surgical revascularization aims must be scheduled for clinically indicated indirect surgical revascularization of at least one hemisphere
4. Speak and read English

Healthy controls

1. No major medical conditions
2. Age = 18-60 years
3. Speak and read English
4. Able to complete 2 study MRIs and all other study procedures

Exclusion Criteria:

-Both moyamoya and healthy controls

1. History of other major neurological conditions (including but not limited to Parkinson's disease, Alzheimer's disease, and Multiple Sclerosis) as confirmed by neuroimaging and neurological evaluation (central adjudication committee).
2. History of traumatic brain injury
3. Independent medical condition expected to lead to death within two years.
4. Condition associated with syndromic moyamoya (including but not limited to sickle cell disease, atherosclerosis, neurofibromatosis, Down syndrome).
5. Severe respiratory illness including but not limited to asthma or chronic obstructive pulmonary disease.

7. Contraindication to 3 Tesla MRI 8. Pregnancy

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with moyamoya disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2029-09-11 (Estimated); Study Completion 2030-09-11 (Estimated)

PRIMARY OUTCOMES:
Revascularization success | 6 years
  The outcome measure will be the number of patients with successful surgical revascularization.

SECONDARY OUTCOMES:
Infarct development | 6 years
  The number of patients with new cerebral infarctions.

CONTACTS AND LOCATIONS:
Overall Officials: Manus J Donahue, MBA, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
This study will not be sharing IPD with other researchers in order to protect participant privacy.